CLINICAL TRIAL: NCT06098248
Title: A Prospective, Multi-centered, Assessor-blinded Clinical Performance Study to Evaluate the Sensitivity and Specificity of the cCeLL-Ex Vivo Device for Intraoperative Brain Tumor Diagnosis.
Brief Title: Evaluation of cCeLL-Ex Vivo Confocal Microscopy for Real-time Brain Tumor Diagnosis
Acronym: cCeLLExvivo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays in specimen recruitment have increased costs and strained resources, risking study validity. To maintain ethical and scientific integrity, the study will be terminated early.
Sponsor: VPIX Medical (Industry)
Collaborators: Unity Health Toronto (Other); Korea University Anam Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: cCell_Ex vivo-01; Republic of Korea (Other: VPIX Medical Inc.)
Record Dates: First submitted 2023-10-05; First posted 2023-10-24 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Benign Brain Tumor; Malignant Brain Tumor
Keywords: Brain Tumor; Brain Tumor Surgery; Cancer Surgery; Brain Tumor Resection; Biopsy; Digital Biopsy; Frozen Section
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: * All enrolled participants were assigned to the same intervention (i.e., cCeLL - Ex vivo), with no separate control group or comparator.
  * The study's primary purpose was to evaluate the diagnostic performance (sensitivity, specificity) of the investigational device in a single cohort of participants undergoing brain tumor resection.
Masking Description: This trial employed an assessor-blinded design. Specifically, the pathologist who interpreted the cCeLL - Ex vivo images had no access to the patient's clinical information, frozen section results, or permanent section results. By ensuring that the individual responsible for cCeLL - Ex vivo image interpretation was blinded to other diagnostic data, the study minimized bias in determining sensitivity and specificity outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients already scheduled for brain tumor surgery (Experimental): Study Arms and Intervention
  This study compares cCeLL - Ex vivo imaging (test) and frozen section histopathology (control) against permanent section histopathology (reference standard).
  * Test Arm: Uses confocal laser fluorescence microscopy (CLFM) for real-time imaging of resected tumor tissues, analyzed by blinded pathologists.
  * Control Arm: Standard H&E-stained frozen section, requiring tissue processing (30-40 min) for intraoperative diagnosis.
  The study evaluates diagnostic accuracy, sensitivity, and specificity of cCeLL - Ex vivo imaging.
  Interventions: Diagnostic Test: cCeLL - Ex vivo

INTERVENTIONS:
Diagnostic Test: cCeLL - Ex vivo — Neoplastic brain tissue biopsied from participant will be visualized, and images will be captured using cCeLL - Ex vivo.

SUMMARY:
Intra-operative evaluation of residual brain tumor currently relies on frozen-section histopathology, which typically requires 20-30 minutes for tissue processing and interpretation, prolonging operative time and increasing staffing demands. Confocal Laser Fluorescence Microscopy (cCeLL - Ex vivo) acquires real-time, high-resolution fluorescence images of resected tissue and therefore may serve as a rapid alternative or adjunct to frozen sections. This prospective, multi-center study was designed to systematically assess the clinical performance of cCeLL - Ex vivo during brain-tumor surgery.

DETAILED DESCRIPTION:
Primary Objective

Demonstrate non-inferiority of cCeLL - Ex vivo versus frozen-section histopathology in terms of clinical sensitivity and specificity for intra-operative brain-tumor diagnosis.

Secondary Objectives Compare diagnostic turnaround time between cCeLL - Ex vivo and frozen section. Evaluate tumor-type classification accuracy for each modality. Determine the average number of images required for definitive cCeLL - Ex vivo interpretation.

Quantify overall diagnostic performance of cCeLL - Ex vivo using the area under the ROC curve (AUC).

ELIGIBILITY:
Inclusion Criteria

Specimens and images used in this study must meet all of the following criteria:

1. Tissue obtained from male or female patients aged 19 years or older.
2. Tissue collected from patients scheduled for neurosurgical resection of a suspected brain tumor.
3. Tissue obtained from patients capable of understanding and signing the informed consent form.

Exclusion Criteria

Specimens and images that meet any of the following criteria will be excluded from the study:

1. Emergency cases where informed consent could not be obtained before surgery.
2. Specimens with significant hemorrhage, affecting image quality.
3. Small biopsy specimens that do not meet the required size for imaging.
4. Poor-quality images that do not meet study criteria, including:

   * Low-quality cCeLL - Ex vivo images.
   * Non-diagnostic cCeLL - Ex vivo images of the tumor core.
5. Cases deemed inappropriate for the study by the principal investigator or study staff due to ethical concerns or potential impact on study results.
6. Patients undergoing multiple surgeries at the same site.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Das, MD,MMSc,PhD, Principal Investigator — Unity Health- St. Michael's Hospital; Shin-Hyuk Kang, MD,MMSc,PhD, Study Director — Korea University
Locations (4):
- St. Michael's Hospital, Toronto, Ontario, Canada
- South Korea (3):
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amos WB, White JG. How the confocal laser scanning microscope entered biological research. Biol Cell. 2003 Sep;95(6):335-42. doi: 10.1016/s0248-4900(03)00078-9. PMID 14519550
- [Background] BIS Research Inc. Medical market data. Updated 2022. https://blog.bisresearch.com/bis-research-market-insights-quick-bytes
- [Background] Carl Zeiss Meditec AG. Convivo: Putting in vivo cellular imaging at your fingertips. 2019:Brochure. Available at: https://www.zeiss.com/content/dam/Meditec/ref_master/products/convivo/documents/convivo_brochure.pdf
- [Background] Chand P, Amit S, Gupta R, Agarwal A. Errors, limitations, and pitfalls in the diagnosis of central and peripheral nervous system lesions in intraoperative cytology and frozen sections. J Cytol. 2016 Apr-Jun;33(2):93-7. doi: 10.4103/0970-9371.182530. PMID 27279685
- [Background] de Martel C, Georges D, Bray F, Ferlay J, Clifford GM. Global burden of cancer attributable to infections in 2018: a worldwide incidence analysis. Lancet Glob Health. 2020 Feb;8(2):e180-e190. doi: 10.1016/S2214-109X(19)30488-7. Epub 2019 Dec 17. PMID 31862245
- [Background] Ferlay J, Ervik M, Lam F, Colombet M, Mery L, Piñeros M, et al. Global Cancer Observatory: Cancer Today. Lyon: International Agency for Research on Cancer; 2020 (https://gco.iarc.fr/today, accessed February 2021).
- [Background] IndustryARC. Oncology Market - Forecast (2020 - 2025). 2020.
- [Background] Mat Zin AA, Zulkarnain S. Diagnostic Accuracy of Cytology Smear and Frozen Section in Glioma. Asian Pac J Cancer Prev. 2019 Feb 26;20(2):321-325. doi: 10.31557/APJCP.2019.20.2.321. PMID 30803189
- [Background] Mauna Kea Technologies. Cellvizio: Real-time in vivo cellular imaging platform. 2021:Brochure. Available at: http://www.cellvizio.net/uploads/media/media_pdf/0001/03/MKT-132-EN-Cellvizio%20Web%20Brochure.pdf
- [Background] MAVIG GmbH. Vivascope: Confocal laser scanning microscopy - In vivo histology for cellular level skin analyses in cosmetic research and dermopharmacy. 2019:Brochure. Available at: https://www.vivascope.de/wp-content/uploads/2019/06/Cosmeticbrochure.pdf
- [Background] Samal S, Kalra R, Sharma J, et al. Comparison between crush/squash cytology and frozen section preparation in intraoperative diagnosis of central nervous system lesions. Oncol J India. 2018;1:25-30.
- [Background] Tofte K, Berger C, Torp SH, Solheim O. The diagnostic properties of frozen sections in suspected intracranial tumors: A study of 578 consecutive cases. Surg Neurol Int. 2014 Dec 3;5:170. doi: 10.4103/2152-7806.146153. eCollection 2014. PMID 25593754
- [Background] White JG, Amos WB, Fordham M. An evaluation of confocal versus conventional imaging of biological structures by fluorescence light microscopy. J Cell Biol. 1987 Jul;105(1):41-8. doi: 10.1083/jcb.105.1.41. PMID 3112165
- [Background] WHO. Assessing national capacity for the prevention and control of noncommunicable diseases: report of the 2019 global survey. Geneva: World Health Organization; 2020.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Status: Completed / Enrolled: 285 patients, 358 specimens, drop-out 36 speciments Study Start: Jan 1, 2023 , Primary y Completion: Nov 27, 2024 First enrollment: Korea: Jan 1, 2023 Canada: Jul 5, 2024 Enrollment ended: Korea: Nov 27, 2024 / Canada: Oct 18, 2024 Analyzed: 322 specimens Study Completion Date (database lock and QC): 31 Dec 2024
Pre-assignment Details: This was a single-group, assessor-blinded study with no randomization or run-in period. Adults (≥19) with suspected brain tumors who consented were enrolled. A total of 285 Patient at four sites (three in Korea, one in Canada) joined; Each could yield up to three specimens, resulting in 322 analyzable samples. No comparator was used, so all proceeded to cCeLL - Ex vivo. No extra screening or washout was performed.
Units Other Than Participants: specimens
Groups:
- Participants: "All participants underwent the same imaging intervention (cCeLL - Ex vivo); Participant Flow counts are reported for both participants and the tissue-specimen units analyzed."
Period: Overall Study
Arm/Group | Participants
Started | 285; 358 specimens
Completed | 271; 322 specimens
Not Completed | 14; 36 specimens

BASELINE CHARACTERISTICS:
Population: The final analyzable dataset consisted of 271 participants(322 specimens)
Units Other Than Participants: Specimens
Groups:
- CeLL - Ex Vivo Imaging: All resected brain-tumor specimens were imaged in the operating room with cCeLL - Ex vivo, a confocal laser fluorescence endomicroscope that captures real-time, sub-cellular resolution images. Blinded expert pathologists interpreted the images on a secure workstation.
Arm/Group | CeLL - Ex Vivo Imaging
Number analyzed (Participants) | 271
Number analyzed (Specimens) | 322
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years at the time of neurosurgical resection, calculated from date of birth. Reported as mean ± SD
  years | 55.6 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth, obtained from medical records. Reported as count and percentage of participants
  Participants
    Female | 154
    Male | 117
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Baseline Number of Tissue Specimens Collected for cCeLL - Ex vivo Imaging [Number; unit: Specimens] | 322

OUTCOME MEASURES:

1. Primary Outcome: Clinical Sensitivity for Tumor Detection (Specimen-level)
Description: The diagnostic results of cCeLL - Ex vivo imaging interpretation by experts and frozen section examination for 283 tumor specimens are presented below.
Time Frame: From neurosurgical resection to permanent pathology (≈ 4 weeks)
Population: Both tumor and non-tumor specimens were collected from 19 participants.
Measure: Number (95% Confidence Interval); unit: Percentage of tumor specimens (%)
Units Other Than Participants: specimens
Groups:
- cCeLL - Ex vivo and Frozen Section: Sensitivity: 256 participants(283 tumor specimens)
Arm/Group | cCeLL - Ex vivo and Frozen Section
Number analyzed (Participants) | 256
Number analyzed (specimens) | 283
Percentage of tumor specimens (%)
  cCeLL - Ex vivo | 96.05 [92.80 to 98.30]
  Frozen section | 94.81 [92.18 to 96.76]
Statistical Analysis 1: Comparison: cCeLL - Ex vivo and Frozen Section; We performed a paired comparison within the same participant population, evaluating both cCeLL - Ex vivo and Frozen Section on each specimen; Test type: Non-Inferiority — The non-inferiority margin was set at 0.05 for sensitivity. A power calculation was conducted assuming a 30% missing data rate, with final missing data at approximately 10%; p < 0.4049, McNemar — A one-sided significance level of 0.05 was used for the non-inferiority tests; McNemar's test was chosen due to paired nominal data (specimens tested by both methods). Degrees of freedom = 1; Risk Difference (RD) = -0.0123, 95% CI 1-sided [upper limit 0.0164], Standard Error of Mean 0.0132 — Lower Limit reflects estimated value due to 1-sided CI requirement and system constraints. True lower bound is theoretically -∞; If any secondary analyses could not fit into the above format (e.g., AUC analysis, time efficiency), they were reported as descriptive statistics rather than hypothesis testing

2. Primary Outcome: Clinical Specificity for Tumor Detection (Specimen-level)
Description: The diagnostic results of cCeLL - Ex vivo imaging interpretation by experts and frozen section examination for 39 normal specimens are as follows
Time Frame: From neurosurgical resection to permanent pathology (≈ 4 weeks)
Population: Both tumor and non-tumor specimens were collected from 19 participants.
Measure: Number (95% Confidence Interval); unit: Percentage of normal specimens (%)
Units Other Than Participants: specimens
Groups:
- cCeLL - Ex vivo and Frozen Section: Specificity: 32 participants(39 normal specimens)
Arm/Group | cCeLL - Ex vivo and Frozen Section
Number analyzed (Participants) | 32
Number analyzed (specimens) | 39
Percentage of normal specimens (%)
  Frozen Section | 67.86 [54.2 to 79.1]
  cCeLL - Ex vivo | 78.57 [65 to 89.9]
Statistical Analysis 1: Comparison: cCeLL - Ex vivo and Frozen Section; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The non-inferiority margin was set at 0.10 for specificity; p < 0.3075, McNemar — A one-sided significance level of 0.10 was used for the non-inferiority tests; McNemar's test was chosen due to paired nominal data (specimens tested by both methods). Degrees of freedom = 1; Risk Difference (RD) = -0.1071, 95% CI 2-sided [-0.1628 to 0.0557], Standard Deviation 0.4103 — [estimate comment as in outcome 1, analysis 1]; f any secondary analyses could not fit into the above format (e.g., AUC analysis, time efficiency), they were reported as descriptive statistics rather than hypothesis testing

ADVERSE EVENTS:
Time Frame: From specimen collection during surgery through final pathology reporting (up to 4 weeks post-surgery)
Description: Adverse events were actively monitored for all 285 participants from specimen collection through final pathology reporting; no adverse events were observed.
Groups:
- Single Group: cCeLL - Ex vivo and Frozen Section: All enrolled participants underwent neurosurgical resection for suspected brain tumors. Resected specimens were examined using the investigational device, cCeLL - Ex vivo (confocal fluorescence endomicroscopy), as well as the standard frozen section procedure. Permanent section served as the final reference standard for comparison.
Arm/Group | Single Group: cCeLL - Ex vivo and Frozen Section
All-Cause Mortality (participants affected / at risk) | 0/285
Serious Adverse Events (participants affected / at risk) | 0/285
Other Adverse Events (participants affected / at risk) | 0/285

LIMITATIONS AND CAVEATS:
1. Ex vivo design restricts immediate in vivo application.
2. Single-arm structure limits certain statistical inferences.
3. Learning curve affects imaging time.
4. Results may not fully generalize beyond the study settings.
5. Some data were missing, though at a low rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT06098248/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT06098248/ICF_001.pdf